CLINICAL TRIAL: NCT00644332
Title: An Open-label, Multi-center Study Evaluating the Validity, Reliability, and Responsiveness of a New Women's Ischemia Symptom Questionnaire in Women With Chronic Angina Treated With Ranolazine Extended-release Tablets (CVT 3041)
Brief Title: An Open-label, Multi-center Study Evaluating the Validity, Reliability, and Responsiveness of a New Female-specific Angina Questionnaire in Women With Chronic Angina Treated With Ranolazine Extended-release Tablets (CVT 3041)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CVT 3041
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Results first posted 2012-07-02 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Angina
MeSH Terms: interventions — Ranolazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ranolazine — Oral dosage form.
  Other Names: Ranexa

SUMMARY:
According to the American Heart Association (AHA) 2011 update of heart disease and stroke statistics, more than 9 million adult patients in the United States (US) have angina. This update also notes that a study of 4 national cross-sectional health examination studies found that, among Americans 40 to 74 years of age, the age-adjusted prevalence of angina was higher among women than men. Per ACC/AHA guidelines, the goal of antianginal therapy is the complete or near complete elimination of anginal chest pain and a return to normal activities and functional capacity. However, evaluating angina and responses to antianginal therapy is often not straightforward. This is particularly true of female patients with angina. Because angina and response to antianginal therapy may differ in men and women, an instrument designed specifically to address symptomatology in women with angina could enhance our understanding and characterization of angina and responses to therapy in this population. The current study will evaluate the validity, reliability, and responsiveness of the newly developed Women's Ischemia Symptom Questionnaire (WISQ) based on changes in angina symptomatology in a female angina population treated with ranolazine, compared with the widely used Seattle Angina Questionnaire (SAQ).

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months of documented history of stable angina or angina equivalents that is relieved by rest and/or sublingual NTG
* Taking antianginal therapy with beta-blockers, and/or dihydropyridine calcium antagonists, and/or long-acting nitrates for at least 4 weeks
* Mean angina frequency of ≥ 2 attacks per week
* Documented clinical evidence of ischemia

Exclusion Criteria:

* Clinically significant hepatic impairment
* Uncontrolled clinically significant cardiac arrhythmias or a history of ventricular fibrillation, torsades de points, or other life-threatening ventricular arrhythmias not associated with acute coronary syndrome
* Treatment with strong cytochrome P450 inhibitors including ketoconazole, itraconazole, clarithromycin, nefazodone, nelfinavir, ritonavir, indinavir, or saquinavir
* Prior treatment with ranolazine
* End-stage renal disease requiring dialysis
* Myocardial infarction or unstable angina

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2007-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nanette K. Wenger, MD, Principal Investigator — Emory University; Noel Bairey Merz, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (28):
- United States (28):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Cardiovascular Consultants, Ltd., Phoenix, Arizona
  - Cardiology Consultants of Orange County, Anaheim, California
  - Access Clinical Trials/Cardiovascular Research Institute (ACT/CVRI), Beverly Hills, California
  - Escondido Cardiology Associates, Escondido, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mission Internal Medical Group, Mission Viejo, California
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Guerra Cardiology, Coral Gables, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - St. Luke Cardiology Associates, Jacksonville, Florida
  - Jacksonville Heart Center, PA, Jacksonville, Florida
  - Emory University & Grady Health System, Atlanta, Georgia
  - Mercy Physician Group Cardiology, Nampa, Idaho
  - North Shore Cardiology, Bannockburn, Illinois
  - Gateway Cardiology, P.C., Jerseyville, Illinois
  - Northern Indiana Research Alliance, Fort Wayne, Indiana
  - Ashland Hospital Corporation d/b/a King's Daughters Medical Center, Ashland, Kentucky
  - University of Louisville, Division of Cardiovascular Medicine, Louisville, Kentucky
  - Gateway Cardiology, P.C., St Louis, Missouri
  - Integrated Cardiology Consultants, LLC d.b.a. Bryan LGH Heart Institute, Lincoln, Nebraska
  - Albany Associates in Cardiology, Albany, New York
  - Total Heart Care, PC, New York, New York
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - St. Vincent Mercy Medical Center, Cardiac Research, Toledo, Ohio
  - BlueStem Cardiology, Bartlesville, Oklahoma
  - Tri-State Medical Group, Cardiology, Sewickley Valley Medical Group, Cardiology, Beaver, Pennsylvania
  - Cardiology Consultants of Philadelphia, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at a total of 30 study sites in the US. The first patient was screened on 07 November 2007, and the last patient was screened on 06 December 2010. The last patient observation was on 20 January 2011.
Pre-assignment Details: In the 2-week qualifying phase, patients continued antianginal medications without changing dose or frequency and completed questionnaires to document angina symptoms, treatment and status. Patients who had average angina frequency of ≥ 2 attacks/week during this phase and met all enrollment criteria were enrolled in the open-label treatment phase.
Groups:
- Ranolazine: In the open-label treatment phase (approximately 4 weeks' duration), patients were given open-label ranolazine extended-release (ER) tablets 500 mg twice daily and continued to take their baseline antianginal medications. Patients completed self-administered questionnaires to document angina symptoms, response to antianginal treatment, and functional status. They also completed daily diaries to document the occurrence of angina episodes and NTG consumption.
Period: Overall Study
Arm/Group | Ranolazine
Started | 171 (172 patients were enrolled; one withdrew consent prior to starting treatment)
Completed | 150
Not Completed | 21
Not completed — Adverse Event | 11
Not completed — Withdrawal by Subject | 6
Not completed — Completion Status Unknown | 2
Not completed — Did Not Meet Eligibility Requirements | 1
Not completed — Could Not Attend Scheduled Visits | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ranolazine
Number analyzed (Participants) | 171
Age Continuous [Mean (Standard Deviation); unit: years] | 64.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3
  Black | 20
  Caucasian | 143
  Hispanic | 5
Region of Enrollment [Number; unit: participants]
  United States | 171
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.5 (6.3)
Weight [Mean (Standard Deviation); unit: kg] | 76.7 (17.6)

OUTCOME MEASURES:

1. Secondary Outcome: Determine Whether the WISQ is Noninferior to the Seattle Angina Questionnaire (SAQ) With Regard to Angina Frequency Items Based on Changes From Baseline (BL) in the Angina Frequency Items of the WISQ With the SAQ Following Ranolazine Treatment
Description: Changes from BL in angina frequency items following ranolazine treatment were measured. Analysis: multiple linear regression; response variable: ΔWISQ - ΔSAQ; independent variables: age and BL WISQ and SAQ scores. WISQ items: 15 points (higher=more severe state); SAQ items: 12 points (lower=more severe state). WISQ scores were recalibrated by multiplying by .75. Noninferiority was to be considered demonstrated if the lower limit of a 2-sided 95% CI for WISQ mean - SAQ mean was above the prespecified margin (WISQ vs SAQ difference of -2).
Time Frame: Baseline to 4 Weeks
Population: Modified Intent-to-Treat Analysis Set
Measure: Number (95% Confidence Interval); unit: ratio of variance
Arm/Group | Ranolazine
Number analyzed (Participants) | 159
ratio of variance | -0.035 [-0.36 to 0.29]

2. Secondary Outcome: Compare Changes From Baseline (BL) in the Physical Limitation Items of the WISQ With the SAQ Following Ranolazine Treatment
Description: Changes from BL in stress, excitement, temperature, satiety, anger, and other limitation items following ranolazine treatment were measured. Analysis: multiple linear regression; response variable: ΔWISQ - ΔSAQ; independent variables: age and BL WISQ and SAQ scores. WISQ items: 27 points (higher=more severe state); SAQ items: 45 points (lower=more severe state). WISQ scores were recalibrated by multiplying by 15/27. Noninferiority was to be considered demonstrated if the lower limit of a 2-sided 95% CI for WISQ mean - SAQ mean was above the prespecified margin (WISQ vs SAQ difference of -2).
Time Frame: Baseline to 4 Weeks
Population: Modified Intent-to-Treat Analysis Set
Measure: Number (95% Confidence Interval); unit: SAQ scale units
Arm/Group | Ranolazine
Number analyzed (Participants) | 159
SAQ scale units | 12.2 [11.3 to 13.2]

3. Secondary Outcome: Compare Changes From Baseline (BL) in Other Like Items of the WISQ With the SAQ Following Ranolazine Treatment
Description: as for outcome 2
Time Frame: Baseline to 4 Weeks
Population: Modified Intent-to-Treat Analysis Set
Measure: Number (95% Confidence Interval); unit: SAQ scale units
Arm/Group | Ranolazine
Number analyzed (Participants) | 159
SAQ scale units | -6.0 [-6.4 to -5.7]

4. Primary Outcome: Evaluate the Validity of the WISQ in Women With Chronic Angina Based on Changes in Patient-reported Angina Frequency and Nitroglycerin (NTG) Consumption Before and Following Treatment With Ranolazine Assessed as Coefficient of Determination (R^2)
Description: Validity of the WISQ was assessed by regression analysis. Results of this analysis are reported as the estimated coefficient of determination (R^2) of the WISQ Total Score at 4 weeks regressed on 4-week angina frequency, 4-week NTG use, and DASI score at 4 weeks. For mean (SEM) Baseline and Week 4 values for angina frequency and NTG use, please refer to Secondary Outcome Measures 7 and 8. For mean (SEM) Baseline and Week 4 DASI values, please refer to Secondary Outcome Measure 9.
Time Frame: Baseline to Week 4
Population: Modified Intent-to-Treat Analysis Set, defined as all patients who took at least 1 dose of ranolazine and completed both baseline and postbaseline questionnaires. Partially missing questionnaire responses were imputed by the methods specified in the scoring instructions; completely missing responses were not imputed.
Measure: Number; unit: coefficient of determination
Arm/Group | Ranolazine
Number analyzed (Participants) | 159
coefficient of determination | 0.337

5. Secondary Outcome: Determine the Effect of Ranolazine on Angina Frequency as Measured by Patient-reported Diaries
Description: Angina episodes were recorded by subjects in their diaries. Weekly frequency of angina episodes was calculated for the two-week baseline period and the last two weeks of the study.
Time Frame: Baseline to Week 4
Population: Modified Intent-to-Treat Analysis Set
  Missing values were excluded
Measure: Mean (Standard Error); unit: attacks per week
Arm/Group | Ranolazine
Number analyzed (Participants) | 154
attacks per week
  Baseline | 7.9 (0.7) [-4.0 to -2.5]
  Week 4 | 3.2 (0.6)
Statistical Analysis 1: Comparison: Ranolazine; Mean change in angina frequency from Baseline to Week 4; Test type: Superiority or Other; Mean Difference (Net) = -4.7, Standard Error of Mean 0.5

6. Secondary Outcome: Determine the Effect of Ranolazine on Nitroglycerin Consumption as Measured by Patient-reported Diaries
Description: Nitroglycerin use was recorded by subjects in their diaries. Weekly frequency of NTG use was calculated for the two-week baseline period and the last two weeks of the study.
Time Frame: Baseline to Week 4
Population: Modified Intent-to-Treat Analysis Set
  Missing values were excluded
Measure: Mean (Standard Error); unit: uses per week
Arm/Group | Ranolazine
Number analyzed (Participants) | 154
uses per week
  Baseline | 4.3 (0.5) [-2.0 to -0.5]
  Week 4 | 1.1 (0.2)
Statistical Analysis 1: Comparison: Ranolazine; Mean change in NTG use from Baseline to Week 4; Test type: Superiority or Other; Mean Difference (Net) = -3.2, Standard Error of Mean 0.5

7. Secondary Outcome: Determine Changes From Baseline in the Duke Activity Status Index (DASI) Following Ranolazine Treatment
Description: The DASI was analyzed as mean values at baseline and Week 4. The DASI is a self-administered questionnaire that measures a patient's functional capacity. It can be used to get a rough estimate of a patient's peak oxygen uptake. The maximum score for the DASI is 58.2 (better functional ability/capacity) and the minimum score is 0 (worse functional ability/capacity).
Time Frame: Baseline to Week 4
Population: Modified Intent-to-Treat Analysis Set
Measure: Mean (Standard Error); unit: DASI scale units
Arm/Group | Ranolazine
Number analyzed (Participants) | 159
DASI scale units
  Baseline | 23.9 (1.1)
  Week 4 | 26.8 (1.1)
Statistical Analysis 1: Comparison: Ranolazine; Test type: Superiority or Other; Mean Difference (Net) = 2.9, Standard Error of Mean 0.8

8. Primary Outcome: Evaluate the Reliability of the WISQ in Women With Chronic Angina Based on Changes in Patient-reported Angina Frequency and NTG Consumption Before and Following Treatment With Ranolazine Assessed as Cronbach's Alpha Value
Description: Reliability of the WISQ was assessed by estimating Cronbach's alpha (standardized); values of 0.7 or higher were to be considered adequate. (Standardized Cronbach's alpha is a coefficient of reliability or consistency, and is a function of the average inter-item correlation.) Cronbach's alpha was calculated for the WISQ instrument overall and for the Angina Frequency/Severity and Angina Stability subscales. Missing item responses were not imputed.
Time Frame: Baseline to Week 4
Population: Modified Intent-to-Treat Analysis Set
Measure: Number; unit: ratio of variances
Arm/Group | Ranolazine
Number analyzed (Participants) | 159
ratio of variances
  WISQ Overall | 0.851
  WISQ Angina Stability | 0.308
  WISQ Angina Frequency | 0.794

9. Primary Outcome: Evaluate the Responsiveness of the WISQ in Women With Chronic Angina Based on Changes in Patient-reported Angina Frequency and NTG Consumption Before and Following Treatment With Ranolazine Assessed by Regression Analysis
Description: Responsiveness of the WISQ was assessed as the estimated coefficient of determination (R^2) of the change from baseline WISQ Total Score at 4 weeks regressed on change from baseline angina frequency and change from baseline NTG use. For mean (SEM) Baseline and Week 4 values for angina frequency and NTG use, please refer to Secondary Outcome Measures 7 and 8.
Time Frame: Baseline to Week 4
Population: Modified Intent-to-Treat Analysis Set
Measure: Number; unit: coefficient of determination
Arm/Group | Ranolazine
Number analyzed (Participants) | 159
coefficient of determination | 0.080

10. Secondary Outcome: Evaluate the Degree of Correlation Between Changes From Baseline in Items of the WISQ and SAQ With Changes From Baseline in Angina Frequency and NTG Diary Data and the DASI
Description: The DASI is a self-administered questionnaire that measures a patient's functional capacity. It can be used to get a rough estimate of a patient's peak oxygen uptake. The maximum score for the DASI is 58.2 (better functional ability/capacity) and the minimum score is 0 (worse functional ability/capacity). The planned analysis was the amount of variation in WISQ and SAQ score changes from baseline explained by changes in angina frequency, NTG use, and DASI score assessed by multiple linear regression analysis.
Time Frame: Baseline to Week 4
Population: Data was collected for this outcome, however, the analysis was not done.
Measure: Number; unit: coefficient of determination
Arm/Group | Ranolazine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Ranolazine
Serious Adverse Events (participants affected / at risk) | 8/171
Other Adverse Events (participants affected / at risk) | 34/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranolazine (N=171)
Acute coronary syndrome (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Chest pain (General disorders) | 3
Non-cardiac chest pain (General disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Pubic rami fracture (Injury, poisoning and procedural complications) | 1
Dizziness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Haematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranolazine (N=171)
Nausea (Gastrointestinal disorders) | 22
Dizziness (Nervous system disorders) | 9
Headache (Nervous system disorders) | 9

LIMITATIONS AND CAVEATS:
The study was terminated early at 86% of targeted enrollment (172 of approximately 200 subjects).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years